CLINICAL TRIAL: NCT01488409
Title: The Effects of Short Term Acipimox Treatment on Skeletal Muscle Phosphocreatine Recovery in Obesity
Brief Title: Effects of Acipimox on Mitochondrial Function in Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-P-000175
Record Dates: First submitted 2011-12-02; First posted 2011-12-08 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Abdominal Obesity; Insulin Resistance; Hypertriglyceridemia
MeSH Terms: conditions — Obesity, Abdominal; Insulin Resistance; Hypertriglyceridemia | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acipimox (Experimental): Treatment with the study drug Acipimox
  Interventions: Drug: Acipimox
- Placebo (Placebo Comparator): Treatment with Placebo control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acipimox — 250 mg by mouth (PO) three times daily
  Arms: Acipimox
Drug: Placebo — 0 mg by mouth (PO) three times daily
  Arms: Placebo

SUMMARY:
The purpose of the study is to examine whether a medication called acipimox can improve your body's mitochondria. Mitochondria are the "power house" of the cell and make energy for your body.

Obesity is associated with increased risk for developing diabetes. However, the investigators do not know how obesity leads to diabetes. Previous studies have shown levels of fat in the blood (free fatty acids or FFA) are higher in obesity, and elevated FFA can affect how our body uses glucose and responds to insulin. Recent studies have shown that changes in mitochondria may be involved in the development of diabetes and may be affected by FFA. The investigators propose to improve the function of mitochondria in obese people with pre-diabetes by treating with acipimox, a medication which decreases FFA. The investigators will use state of the art techniques to evaluate the mitochondria, including a new magnetic resonance imaging (MRI) technique to measure function of mitochondria in muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-55 years old
2. Body Mass Index (BMI) ≥ 30 kg/m2
3. Waist circumference ≥ 102 cm in men and ≥ 88 cm in women
4. Hypertriglyceridemia defined as triglycerides ≥ 150 mg/dl OR Insulin resistance defined as elevated fasting glucose (≥ 100 mg/dl but <125 mg/dl) or hyperinsulinemia defined as fasting serum insulin ≥ 10 uU/ml.

Exclusion Criteria:

1. Subjects on any hormonal treatment including estrogen, hormone replacement therapy, oral contraceptives, testosterone, glucocorticoids, anabolic steroids, GH, GH releasing hormone or Insulin like growth factor (IGF)-1 within 3months of enrollment.
2. Subjects who have a known history of diabetes, using any anti-diabetic drugs, or fasting blood glucose of ≥ 125 mg/dl.
3. Use of cholesterol lowering medication including niacin or fish oil.
4. Changes in anti-hypertensive regimen within 3months of screening.
5. Chronic illness including HIV, anemia (Hgb <12 g/dL), chronic kidney disease (Creatinine > 2 mg/dL), or liver disease (SGOT > 2.5 x upper limit normal).
6. Use of Aspirin, Clopidogrel (Plavix), Warfarin (Coumadin) or other anti-coagulants
7. History of or active peptic ulcer disease
8. History of any recent cardiovascular event including myocardial infarction (MI; heart attack), cerebral vascular accident (CVA; or stroke) or transient ischemic attack (TIA; or mini-stroke) within 3 months of screening visit, unstable angina pectoris, oxygen-dependent severe pulmonary disease
9. Subjects with contraindication for an MRI study including any significant metal in their body including surgical clippings, or pacemakers and known claustrophobia.
10. History of recent alcohol or substance abuse (< 1 year)
11. Positive pregnancy test or lactating females
12. Women of child-bearing potential not currently using non-hormonal birth control methods including barrier methods (intra-uterine device or IUD, condoms, diaphragms) or abstinence
13. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Makimura H, Stanley TL, Suresh C, De Sousa-Coelho AL, Frontera WR, Syu S, Braun LR, Looby SE, Feldpausch MN, Torriani M, Lee H, Patti ME, Grinspoon SK. Metabolic Effects of Long-Term Reduction in Free Fatty Acids With Acipimox in Obesity: A Randomized Trial. J Clin Endocrinol Metab. 2016 Mar;101(3):1123-33. doi: 10.1210/jc.2015-3696. Epub 2015 Dec 21. PMID 26691888

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acipimox | Placebo
Started | 20 | 19
Completed | 16 | 15
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acipimox | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (5) | 45 (7) | 46 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8 | 10 | 18
  Black | 12 | 8 | 20
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Phosphocreatine Recovery (ViPCr) at 6-months
Description: The rate of recovery of phosphocreatine concentration after depletion by exercise is considered a measurement of mitochondrial function. Change in phosphocreatine recovery from baseline to 6 months will therefore give a measurement of change in mitochondrial function. ViPCR is given -- a higher value indicates better mitochondrial function.
Time Frame: Change from Baseline to 6-months Visit
Population: all available data used
Measure: Mean (Standard Deviation); unit: mM/s
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 16 | 12
mM/s | 1.7 (9.6) | 1.6 (10.8)
Statistical Analysis 1: Comparison: Acipimox vs Placebo; Test type: Superiority or Other; p = 0.97, t-test, 2 sided

2. Secondary Outcome: Change From Baseline in Insulin Sensitivity at 6-months
Description: Change in insulin resistance assessed by hyperinsulinemic-euglycemic clamp study at Baseline and at 6-months. Change in insulin-stimulated glucose uptake (M) during 40 mU/m2/min insulin clamp is given.
Time Frame: Change from Baseline to 6-months visit
Population: all available data used
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 15 | 14
mg/kg/min | 0.1 (1.9) | 0.2 (1.4)
Statistical Analysis 1: Comparison: Acipimox vs Placebo; Test type: Superiority or Other; p = 0.85, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Mitochondrial Density at 6 Months
Description: Muscle tissue obtained from biopsy will be used to assess mitochondrial number and morphology by microscopes at Baseline and at 6-months. The change in mitochondrial density from 6 months to baseline is given.
Time Frame: Change from Baseline to 6-months
Population: all available data used
Measure: Mean (Standard Deviation); unit: percentage of total muscle fiber area
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 8 | 9
percentage of total muscle fiber area | 0.4 (1.3) | 0 (1.6)
Statistical Analysis 1: Comparison: Acipimox vs Placebo; Test type: Superiority or Other; p = 0.52, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Intramyocellular Lipid Content at 6-months
Description: Change in tibialis intramyocellular lipid (IMCL) normalized to creatinine is given.
Time Frame: Change from Baseline to 6-months
Population: all available data used
Measure: Mean (Standard Deviation); unit: ratio of IMCL peak to Creatinine peak
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 14 | 15
ratio of IMCL peak to Creatinine peak | -0.2 (3.0) | 0.0 (2.3)
Statistical Analysis 1: Comparison: Acipimox vs Placebo; Test type: Superiority or Other; p = 0.79, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Lipid Profile at 6-months
Description: Change in direct low density lipoprotein (LDL) cholesterol is given
Time Frame: Change from Baseline to 6-months
Population: all available data used
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 16 | 15
mg/dL | -19 (26) | 6 (22)
Statistical Analysis 1: Comparison: Acipimox vs Placebo; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Acipimox | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 16/20 | 16/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acipimox (N=20) | Placebo (N=19)
Flushing (Skin and subcutaneous tissue disorders) | 8 | 4
nausea (Gastrointestinal disorders) | 4 | 3
Dizziness (General disorders) | 1 | 1
abdominal bloating (Gastrointestinal disorders) | 3 | 2
dry mouth (General disorders) | 1 | 0
gastroesophageal reflux (Gastrointestinal disorders) | 7 | 5
pain following biopsy (Surgical and medical procedures) | 0 | 1
bleeding following biopsy (Surgical and medical procedures) | 1 | 1
abdominal pain (Gastrointestinal disorders) | 2 | 2
diarrhea (Gastrointestinal disorders) | 7 | 2
vomiting (Gastrointestinal disorders) | 0 | 1
joint pain and swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 1 | 0
loss of appetite (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No